CLINICAL TRIAL: NCT01342185
Title: A Randomized, Controlled, Open-label, Multicenter Clinical Study of Treatment of Chronic Hepatitis B With TY-CZ-9999 Ozone Therapy System
Brief Title: Efficacy of Medical Ozone Therapy in Patients With Chronic Hepatitis B
Acronym: EMOTCHB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Tianyi medical instruments limited company, Ningbo, China (Unknown)
Responsible Party: Principal Investigator, guoyabing, professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: a4xr2dv8
Record Dates: First submitted 2011-02-16; First posted 2011-04-27 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Hepatitis B
Keywords: Medical ozone therapy; chronic hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Glycyrrhizic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Medical ozone therapy with tianyi (Experimental)
  Interventions: Device: medical ozone therapy with tianyi
- medical ozone therapy with humares (Active Comparator)
  Interventions: Device: medical ozone therapy with humares
- Diammonium glycyrrhizinate Capsules (Placebo Comparator)
  Interventions: Drug: Diammonium glycyrrhizinate Capsules

INTERVENTIONS:
Device: medical ozone therapy with tianyi — Medical ozone therapy with instrument made in China Patients in this arm will receive autohemotherapy. First month: ozone concentration: 20µg ~40µg /ml;The second month: 30µg/ml × 100ml oxygen- ozone gas × 100 ml blood;The third month: 20µg/ml × 100ml oxygen- ozone gas× 100 ml blood.
  Other Names: ozone instrument made in China: TianYi
  Arms: Medical ozone therapy with tianyi
Device: medical ozone therapy with humares — Medical ozone therapy with instrument made in Germany Patients in this group will receive autohemotherapy treatment, regime as ArmⅠ.
  Other Names: ozone instrument made in Germany: Humares
  Arms: medical ozone therapy with humares
Drug: Diammonium glycyrrhizinate Capsules — Drug: Diammonium glycyrrhizinate Capsules Patients in this group will receive oral Diammonium glycyrrhizinate Capsules 150mg, three times a day for 12 weeks.
  Other Names: ganlixin capsules
  Arms: Diammonium glycyrrhizinate Capsules

SUMMARY:
The purpose of this study is to verify the effectiveness and safety of medical ozone therapy system in treatment of chronic hepatitis B.

DETAILED DESCRIPTION:
Total of 189 patients with compensated chronic hepatitis B will be divided equally and randomly into three arms. Patients in arm I and II treated with medical ozone therapy with different medical ozone generators, one was made in Tianyi medical instruments limited company and the other in Germany. Sixty-three patients of arm III treated with Diammonium glycyrrhizinate Capsules, common used liver protective herb drug. The term of therapy is 12 weeks. Virology response, biochemistry response and hepatitis B viral serological response will be studied at the end of 12 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, not less than 16 years old；
2. HBsAg positive for over 6 months；
3. ALT over 2×ULN, TBIL less than 80µmol/L and serum HBV DNA over 10000copies/ml。

Exclusion Criteria:

1. Patient has a history of hemorrhagic or hemolysis disease;
2. Patient has any history of clinical signs/symptoms of hepatic decompensation or serious metabolic hepatic disease;
3. Patient is co-infected with HIV or HCV;
4. Patient is treated with anti-virus drug like interferon or nucleoside analogue in recent 6 months;
5. Patient is treated with immunosuppressive agent for long time, including patient has a history of organ transplantation;
6. Pregnancy;
7. Current alcohol or drug abuse;
8. Difficulty to draw blood through veins;
9. Patient has a history of carcinoma, or finding suggestive of possible hepatocellular carcinoma (HCC), or AFP over than 100ng/ml;
10. Patient has a history of any severe physical disease such as cardio-vascular, kidney events, hyperthyroidism or serious electrolyte disturbance;
11. Patient is enrolled in any other clinical trials.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
HBV DNA | week 12
  To demonstrate the percentage of patients achieving HBV DNA<1000copies/mL or decreased 100 times at week 12.

SECONDARY OUTCOMES:
HBeAg | week12
  Percentage of patients with HBeAg loss and HBeAg seroconversion at week 12 in patients with HBeAg positive at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: yabing guo, professor, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China